CLINICAL TRIAL: NCT02086253
Title: Role of Endothelin-1 in Mediating Flow-mediated Dilatation of Conduit Arteries During Sustained Hyperemic Stimulation
Brief Title: Role of Endothelin-1 in Flow-mediated Dilatation
Acronym: Endothelin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 2013/161/HP; 2013-004425-87 (EudraCT Number)
Record Dates: First submitted 2014-02-18; First posted 2014-03-13 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Healthy Conditions
Keywords: Endothelin, endothelium, flow-mediated dilatation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- BQ-788 (Experimental): Effect of BQ-788 on the magnitude of sustained flow-mediated dilatation
  Interventions: Drug: BQ-788 and/or BQ-123
- BQ-123 (Experimental): Effect of BQ-123 on the magnitude of sustained flow-mediated dilatation
  Interventions: Drug: BQ-788 and/or BQ-123
- BQ-788 + BQ-123 (Experimental): Effect of BQ-788+BQ-123 on the magnitude of sustained flow-mediated dilatation
  Interventions: Drug: BQ-788 and/or BQ-123

INTERVENTIONS:
Drug: BQ-788 and/or BQ-123

SUMMARY:
Endothelial dysfunction of conduit arteries contributes to the increased morbidity and cardiovascular mortality in patients with essential hypertension and appears increasingly as an independent therapeutic target. We have shown previously that besides a decrease in the availability of NO and other endothelium-derived vasodilators factors, the epoxyeicosatrienoic acids, an increase in the vasoconstrictor endothelin-1 (ET-1) may play a role in the pathophysiology of this endothelial dysfunction. Indeed, the local concentrations of endothelin-1 during the endothelium-dependent dilation of the radial artery in response to a sustained increase in blood flow decreased significantly in healthy volunteers controls but not in hypertensive patients. This lack of adaptation of the endothelinergic system could be due to a decreased clearance of endothelin-1 by endothelial ETB receptors, potentiating the vasoconstrictor action of endothelin-1 mediated by ETA receptor activation at the muscular level. However, to validate this hypothesis , it is needed to demonstrate the physiological role of ETA receptor and ETB in sustained flow-mediated dilatation of conduit arteries.

ELIGIBILITY:
Inclusion Criteria:

* Male, Caucasian, aged 18 to 35 years
* Non-Smoking
* Resting heart rate> 50 and <90 bpm
* SBP <140 mmHg and DBP <90 mm Hg at rest in the supine position for 10 minutes
* Normal ECG

Exclusion Criteria:

* Known allergy
* Intolerance to glyceryl trinitrate
* Intolerance to lidocaine
* Family history of hypertension
* Excessive alcohol consumption ( more than 50 g / day)
* Addiction or presumption of illicit drug use
* Subject refusing blood samples for serology of hepatitis B , C and HIV
* History of illness or psychological or sensory abnormality that may prevent the subject to understand the requirements for participation in the protocol or prevents giving informed consent
* Metabolic or endocrine disease
* Immunological diseases
* Renal or hepatic impairment
* Ischemic or obstructive heart disease
* Neoplastic disease
* Gastrointestinal disease
* Neurological disease , intracranial hypertension , seizure disorders
* Compulsive overeating , bulimia, anorexia
* Severe psychiatric illness
* Presence of a clinically significant abnormality in laboratory tests carried out at the inclusion visit .
* HBs Ag , HCV Ab , Ac HIV 1 or HIV 2 positive .
* The use of any drug in the range of less than 5 half-life time, in particular betablockers, sildenafil, cimetidine, amiodarone .

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2014-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Effect of ETB receptor blockade on flow-mediated dilatation | One hour after BQ-788 brachial infusion
  This study will evaluate the effect of the ETB receptor blockade on the magnitude of the flow-mediated dilatation of the radial artery in response to distal skin heating in 8 healthy subjects. Radial artery diameter and blood flow will be measured by high-resolution echotracking coupled to Doppler.

SECONDARY OUTCOMES:
Effect of ETA and ETA/ETB receptor blockade on flow-mediated dilatation | One hour after BQ-123 alone or with BQ-788 brachial infusion
  This study will evaluate the effect of ETA receptor and combined ETA/ETB receptor blockade on the magnitude of the flow-mediated dilatation of the radial artery in response to distal skin heating in 8 healthy subjects. Radial artery diameter and blood flow will be measured by high-resolution echotracking coupled to Doppler.
Effect of ETA and/or ETB receptor blockade on ET-1, NO and EET bioavailability | One hour after BQ-788 and/or BQ-123 brachial infusion
  This study will evaluate the effect of ETA and/or ETB blockade on the variations in the local concentrations of ET-1, NO and EETs during sustained flow-mediated dilation in 8 healthy subjects. For this purpose, local blood samples will be drawn before (34°C) and at the end of hand skin heating (44°C). Plasma nitrite, indicator of NO availability will be quantified by chemiluminescence.Plasma EETs will be quantified by LC-MS. Plasma ET-1 will be quantified with an immunoassay.

CONTACTS AND LOCATIONS:
Overall Officials: Robinson JOANNIDES, Doctor, Principal Investigator — Chu - Hôpitaux de Rouen
Locations (1):
- CHU - Hôpitaux de Rouen, Rouen, Normandy, France